CLINICAL TRIAL: NCT06727760
Title: Investigation of the Effects of Colic Massage and Kangaroo Care on Colicky Infants and Their Mothers
Brief Title: The Effect of Colic Massage and Kangaroo Care on Babies and Their Mothers
Acronym: randomized
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsah Sunay Ertem (Other)
Responsible Party: Sponsor-Investigator, Gulsah Sunay Ertem, Principal Investigator, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-25691463-900-35292
Record Dates: First submitted 2024-11-23; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Colic, Infantile; Crying Time in Colicky Infants; Postpartum Depression; Postpartum Anxiety; Motherhood
Keywords: colic; cangroo care; crying and sleeping duration; nursing education; postpartum anxiety; postpartum depression
MeSH Terms: conditions — Colic; Depression, Postpartum; Crying | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- massage group (Experimental): Colic massage is applied to babies with infantile colic
  Interventions: Behavioral: massage
- kangaroo care group (Experimental): Kangaroo care is applied to babies with infantile colic
  Interventions: Behavioral: kangroo care
- control group (No Intervention): No intervention is applied to babies with infantile colic

INTERVENTIONS:
Behavioral: massage — The mothers in the massage group applied colic massage according to the "Educational Colic Massage Checklist" twice a day for 15-20 minutes each time for three weeks, when the baby was calm and during colic attacks.
  Arms: massage group
Behavioral: kangroo care — The mothers in the kangaroo care group applied kangaroo care according to the "Educational Kangaroo Care Checklist" twice a day for three weeks for 15-20 minutes each time when the baby was calm and during colic attacks.
  Arms: kangaroo care group

SUMMARY:
Background: Infantile colic is a condition characterized by inconsolable crying in infants under three months of age.

Purpose: The aim of this study is to determine the effects of colic massage and kangaroo care on infantile colic symptoms, crying, and sleep duration.

Method: Our study was conducted at the Child Health and Diseases Polyclinic of Atatürk city Hospital between March 2022 and April 2023. The study sample consisted of infants diagnosed with infantile colic who applied to the polyclinic and their mothers. 96 infants were randomly selected in our study using the randomization method. They were assigned to the massage, kangaroo care, and control groups. Infants in the colic massage and kangaroo care groups received interventions for 15-20 minutes in the morning and evening, while the control group received no intervention. Before the intervention, crying and sleep duration were monitored and recorded for 24 hours for one week in all three groups. Mothers continued the massage and kangaroo care application for 3 weeks. In the 3rd week of the application, 24-hour crying and sleep duration were recorded again for one week. Before and after the interventions, the Infantile Colic Scale (ICS) was applied to all three groups. The three groups were compared with the Wilcoxon test.

DETAILED DESCRIPTION:
Data were collected from volunteer mothers of babies diagnosed with infantile colic who applied to the Child Health and Diseases outpatient clinic between March 2022 and February 2023 and who met the inclusion criteria for the study. The mothers were informed about the research through the "Informed Consent Form". Data were collected by the researcher through face-to-face interviews. The "Mother-Baby Information Form", "Infant Colic Scale", "Postpartum Specific Anxiety Scale", "Barkin Maternal Function Scale" and "Beck Depression Scale" were applied to the mothers in the massage, kangaroo care and control groups in the outpatient clinic before the intervention. They were then given the "Crying and Sleep Duration Form" and asked to fill it out at home for a week. Mothers who filled out the crying and sleep duration forms for a week were given an appointment for a home visit. The homes of these mothers were visited and the crying and sleep duration forms filled out for a week were collected. After collection, mothers were taught infantile colic massage and kangaroo care on a baby manikin according to randomization and were allowed to practice (The researcher has a "holistic infant massage certificate"). Mothers in the massage group applied colic massage according to the "Educational Colic Massage Checklist" for 15-20 minutes twice a day for three weeks when the baby was calm and during colic attacks. Mothers in the kangaroo care group applied kangaroo care according to the "Educational Kangaroo Care Checklist" for 15-20 minutes twice a day for three weeks when the baby was calm and during colic attacks. No intervention was made to the mothers in the control group. Mothers in all three groups filled out the "Crying and Sleep Duration Form" again for one week in the last week of the study. At the end of the study, the "Infantile Colic Scale", "Postpartum Specific Anxiety Scale", "Barkin Maternal Function Scale" and "Beck Depression Scale" were applied to the mothers in all three groups again (Mothers were supported with video calls and video recordings during the first massage and kangaroo care application and when needed). The study lasted four weeks in total and the intervention lasted three weeks.

ELIGIBILITY:
Baby's Inclusion Criteria:

* Diagnosed with infantile colic
* Being born at term

Baby's Exclusion Criteria:

* Lactose allergy,
* Diagnosed with another chronic disease
* Skin problem,
* Weighing less than 2500 grams
* Having congenital anomalies
* Vomiting, constipation and malnutrition

Mothers' inclusion criteria

* being a volunteer
* being literate and
* having a smart phone.

Mothers' exclusion criteria

* using incorrect massage and kangaroo care
* using other traditional and medical treatments during the study.

Ages: 3 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
infantile scale scores | up to 3 weeks
  The Infantile Colic Scale consists of 19 questions. The scale has 5 subscales: Cow's Milk/Soy Protein Allergy/Intolerance, Immature Gastrointestinal System, Immature Central Nervous System, Difficult Infant Temperament, Parent-Infant Interaction, and Problematic Infant. Scale items are rated on a Likert-type scale ranging from 1 to 6. Ratings range from 1 (strongly disagree) to 6 (strongly agree). Negative questions were reverse-coded for interpreting the scores. Item 3 in the immature gastrointestinal system subscale, items 7, 8, and 9 in the immature central nervous system subscale, items 13, 14, and 15 in the difficult infant temperament subscale, and items 17 and 19 in the parent-infant interaction and problematic infant subscales were reverse-coded.Data are expressed as mean ± SD and median (minimum: maximum).
mothers' postpartum anxiety scores | up to 3 weeks
  The Postpartum Specific Anxiety Inventory consists of 51 items. Responses to the items are rated on a 4-point Likert scale ranging from 1 to 4 (1=never, 2=sometimes, 3=usually, 4=always). The total score for the level of postpartum anxiety is; below 73 points is considered low risk, between 74 and 100 points is considered moderate risk, and above 101 points is considered high risk. The lowest possible score is 51, and the highest score is 204. 8 The scale has four subscales: Items 1-15 assess maternal adequacy and attachment concerns, items 16-26 assess infant safety and well-being concerns, items 27-33 assess practical infant care concerns, and items 34-51 assess psychosocial adjustment to motherhood.
mother's depression scores | up to 3 weeks
  The scale consists of 21 items related to depressive symptoms such as pessimism, sense of failure, dissatisfaction, guilt, restlessness, fatigue, decreased appetite, indecisiveness, sleep disorders, and social withdrawal. The total score that can be obtained from the scale varies between 0-63. Those who scored 17 and above were accepted as 'depressive symptoms' as 10. The Turkish validity and reliability studies of the BDI were conducted by Teğin in 1980 and by Hisli in 1989, and the Cronbach alpha value was found to be 0.80. The BDI scoring for the severity of depression is interpreted as 0-9 = Minimal, 10-16 = Mild, 17-29 = Moderate, 30-63 = severe, depression. It takes approximately 15 minutes to complete the scale. However, this time may vary depending on the patient's level of education and whether or not they have obsessive characteristics.

SECONDARY OUTCOMES:
maternal function scores. | up to 3 weeks
  The scale's self-care dimension was calculated as 0.66, maternal psychology sub-dimension as 0.71, baby care sub-dimension as 0.62, social support sub-dimension as 0.69, and adaptation to motherhood sub-dimension as 0.50. The responses on the scale are numbered from 0 to 6. 0 is expressed as "completely disagree", 1 as "disagree", 2 as "somewhat disagree", 3 as "undecided", 4 as "somewhat agree", 5 as "agree", and 6 as "completely agree". The lowest score that can be obtained in the scoring of the scale is 0, and the highest score is 96. It is accepted that the functional status increases as the scores increase. BAFÖ is applied to mothers with babies younger than 18 months.
colic babies crying and sleeping time | up to 3 weeks
  It is a form created by the researcher in which infants' daily crying and sleep durations can be recorded at every hour of the day and on every day of the week.

CONTACTS AND LOCATIONS:
Overall Officials: nurcan özyazıcıoğlu, professor, Study Director — bursa uludağ üniversitesi
Locations (1):
- Ataturk City Hospital, Balıkesir, Altıeylül, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Higgins M, St James Roberts I, Glover V. Postnatal depression and mother and infant outcomes after infant massage. J Affect Disord. 2008 Jul;109(1-2):189-92. doi: 10.1016/j.jad.2007.10.027. Epub 2007 Dec 20. PMID 18086500
- [Background] Onozawa K, Glover V, Adams D, Modi N, Kumar RC. Infant massage improves mother-infant interaction for mothers with postnatal depression. J Affect Disord. 2001 Mar;63(1-3):201-7. doi: 10.1016/s0165-0327(00)00198-1. PMID 11246096
- [Background] Lotfalipour B, Tirgari B, Pouraboli B, Mirzaee M. Effect of Preterm Infant Massage by the Mother on the Mood of Mothers Having Preterm Infants. J Chiropr Med. 2019 Mar;18(1):67-76. doi: 10.1016/j.jcm.2018.11.001. Epub 2019 May 7. French. PMID 31193199
- [Background] Lonstein JS. Regulation of anxiety during the postpartum period. Front Neuroendocrinol. 2007 Aug-Sep;28(2-3):115-41. doi: 10.1016/j.yfrne.2007.05.002. Epub 2007 Jun 2. PMID 17604088
- [Background] Lee SB, Shin HS. [Effects of Kangaroo Care on anxiety, maternal role confidence, and maternal infant attachment of mothers who delivered preterm infants]. Taehan Kanho Hakhoe Chi. 2007 Oct;37(6):949-56. doi: 10.4040/jkan.2007.37.6.949. Korean. PMID 17992067
- [Background] Fujita M, Endoh Y, Saimon N, Yamaguchi S. Effect of massaging babies on mothers: pilot study on the changes in mood states and salivary cortisol level. Complement Ther Clin Pract. 2006 Aug;12(3):181-5. doi: 10.1016/j.ctcp.2006.01.003. Epub 2006 Mar 13. PMID 16835028
- [Background] Feijo L, Hernandez-Reif M, Field T, Burns W, Valley-Gray S, Simco E. Mothers' depressed mood and anxiety levels are reduced after massaging their preterm infants. Infant Behav Dev. 2006 Jul;29(3):476-80. doi: 10.1016/j.infbeh.2006.02.003. Epub 2006 Mar 27. PMID 17138300
- [Background] Erduran B, Yaman Sozbir S. Effects of intermittent kangaroo care on maternal attachment, postpartum depression of mothers with preterm infants. J Reprod Infant Psychol. 2023 Nov;41(5):556-565. doi: 10.1080/02646838.2022.2035703. Epub 2022 Feb 7. PMID 35129000
- [Background] Badiee Z, Faramarzi S, MiriZadeh T. The effect of kangaroo mother care on mental health of mothers with low birth weight infants. Adv Biomed Res. 2014 Oct 20;3:214. doi: 10.4103/2277-9175.143262. eCollection 2014. PMID 25371871
- [Background] Anwar F, Warsi A, Ahmed J, Zaidi B, Turab A, Khan MA, Khan KS. The effectiveness of kangaroo mother care in lowering postpartum depression in mothers of preterm and low birth weight babies: a systematic review and meta-analysis. Ann Med Surg (Lond). 2023 Apr 12;85(6):2841-2848. doi: 10.1097/MS9.0000000000000480. eCollection 2023 Jun. PMID 37941566
- [Background] Parsa P, Karimi S, Basiri B, Roshanaei G. The effect of kangaroo mother care on physiological parameters of premature infants in Hamadan City, Iran. Pan Afr Med J. 2018 May 31;30:89. doi: 10.11604/pamj.2018.30.89.14428. eCollection 2018. PMID 30344873
- [Background] Johnson JD, Cocker K, Chang E. Infantile Colic: Recognition and Treatment. Am Fam Physician. 2015 Oct 1;92(7):577-82. PMID 26447441
- [Background] Daelemans S, Peeters L, Hauser B, Vandenplas Y. Recent advances in understanding and managing infantile colic. F1000Res. 2018 Sep 7;7:F1000 Faculty Rev-1426. doi: 10.12688/f1000research.14940.1. eCollection 2018. PMID 30271572
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Background] Zeevenhooven J, Koppen IJ, Benninga MA. The New Rome IV Criteria for Functional Gastrointestinal Disorders in Infants and Toddlers. Pediatr Gastroenterol Hepatol Nutr. 2017 Mar;20(1):1-13. doi: 10.5223/pghn.2017.20.1.1. Epub 2017 Mar 27. PMID 28401050
- [Background] Wolke D, Bilgin A, Samara M. Systematic Review and Meta-Analysis: Fussing and Crying Durations and Prevalence of Colic in Infants. J Pediatr. 2017 Jun;185:55-61.e4. doi: 10.1016/j.jpeds.2017.02.020. Epub 2017 Apr 3. PMID 28385295
- [Background] Sheidaei A, Abadi A, Zayeri F, Nahidi F, Gazerani N, Mansouri A. The effectiveness of massage therapy in the treatment of infantile colic symptoms: A randomized controlled trial. Med J Islam Repub Iran. 2016 Apr 9;30:351. eCollection 2016. PMID 27453882
- [Background] Tekgunduz KS, Gurol A, Apay SE, Caner I. Effect of abdomen massage for prevention of feeding intolerance in preterm infants. Ital J Pediatr. 2014 Nov 14;40:89. doi: 10.1186/s13052-014-0089-z. PMID 25394549
- [Background] Mansouri S, Kazemi I, Baghestani AR, Zayeri F, Nahidi F, Gazerani N. A placebo-controlled clinical trial to evaluate the effectiveness of massaging on infantile colic using a random-effects joint model. Pediatric Health Med Ther. 2018 Nov 16;9:157-163. doi: 10.2147/PHMT.S185214. eCollection 2018. PMID 30532613
- [Background] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Derived] Ertem GS, Ozyazicioglu N. Effects of colic massage and kangaroo care on infantile colic pain, crying and sleep duration: A randomized controlled trial. J Pediatr Nurs. 2025 Sep-Oct;84:390-396. doi: 10.1016/j.pedn.2025.07.003. Epub 2025 Jul 10. PMID 40644765
- See also: Meta-analysis the effect of baby massage in increasing quality of sleep and infant body weight. — https://doi.org/10.26911/thejmch.2024.09.01.05
- See also: The Effects of Kangaroo Mother Care (KMC) on the Fuss and Crying Time of Colicky Infants. Iranian Journal of Neonatology, 6(1). — https://doi.org/10.22038/ijn.2015.4152
- See also: Effects of abdominal massage on feeding tolerance in preterm infants hospitalized in selected hospitals of Isfahan-Iran. — https://doi.org/10.22038/ijp.2017.21376.1795
- See also: Kangaroo Mother Care and Neonatal Outcomes in the Pediatric Department of CHU Gabriel Toure — https://doi.org/10.4236/ojped.2022.121019
- See also: Akdoğan R. The Effect of Spa and Massage Applied to Babies on Colic Symptoms: A Randomized Controlled Trial. PhD Thesis. Istanbul University. Istanbul. 2023 — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Meta-analysis the effect of baby massage in increasing quality of sleep and infant body weight — https://doi.org/10.26911/thejmch.2022.07.01.07
- See also: A controlled trial of skin-to-skin contact in extremely preterm infants. — https://doi.org/10.1016/j.earlhumdev.2005.11.008
- See also: Efficacy of abdominal massage on feeding intolerance of preterm neonetes — https://scholar.google.com.tr/scholar?q=Efficacy+of+abdominal+massage+on+feeding+intolerance+of+preterm+neonates.&hl=tr&as_sdt=0&as_vis=1&oi=scholart
- See also: The effects of infant massage on maternal postpartum depression: A randomized controlled trial. — https://doi.org/10.4103/nms.nms_80_17
- See also: The effects of infant massage on maternal distress: a systematic review — http://dx.doi.org/10.4236/psych.2015.616204
- See also: Comparing the effect of kangaroo mother care and massage on preterm infant pain score, stress, anxiety, depression, and stress coping strategies of their mothers. — https://doi.org/10.22038/ijp.2020.50006.3990
- See also: The impact of baby massage training on awareness, perceived stress and breastfeeding self-efficacy of mothers with hospitalized neonate — https://doi.org/10.22038/ijp.2018.32043.2833
- See also: Infant massage improves attitudes toward childbearing, maternal satisfaction and pleasure in parenting — https://doi.org/10.1016/j.infbeh.2017.08.006
- Available data/document: article: Survey in efficacy of probioti — https://pejouhesh.sbmu.ac.ir/article-1-1582-en.html
- Available data/document: article: Effectiveness of massage — https://scholar.google.com.tr/scholar?q=Effectiveness+of+massage+therapy+for+treatment+of+infantile+colic.&hl=tr&as_sdt=0&as_vis=1&oi=scholart
- Available data/document: article: The effect of massage — https://tumj.tums.ac.ir/browse.php?a_id=11133&slc_lang=en&sid=1&printcase=1&hbnr=1&hmb=1
- Available data/document: rewiev: 0-1 Yaş Arası Bebekler — https://dergipark.org.tr/tr/pub/firattip/issue/6338/84544
- Available data/document: Guide: kangroo care guide — https://www.who.int/publications/i/item/9241590351
- Available data/document: article: The Effects of Kangaroo Mother — https://ijn.mums.ac.ir/article_4152.html
- Available data/document: article: efficacy of probiotic — https://pejouhesh.sbmu.ac.ir/article-1-1582-en.html
- Available data/document: article: Effect of massage — https://scholar.google.com.tr/scholar?q=Effectiveness+of+massage+therapy+for+treatment+of+infantile+colic.&hl=tr&as_sdt=0&as_vis=1&oi=scholart
- Available data/document: doctora thesis: The Effect of Aromatherapy — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp